CLINICAL TRIAL: NCT02066974
Title: Circulating Tumor Cell Genome in Peripheral Blood From Hepatocellular Carcinoma Patients Under Radiotherapy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Shang-Wen Chen, Department of Radiation Oncology, China Medical University, China
Other Study IDs: CMUH102-REC2-112
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Circulating Neoplastic Cells; Adverse Effect of Radiation Therapy; Fatal Outcome
Keywords: hepatocellular carcinoma; genomic expression; radiotherapy
MeSH Terms: conditions — Neoplastic Cells, Circulating; Radiation Injuries; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Fragmented DNA and RNA, Methylation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatoma, Circulating tumor genome: Hepatoma requiring radiotherapy
  Interventions: Genetic: hepatoma requiring radiotherapy

INTERVENTIONS:
Genetic: hepatoma requiring radiotherapy — hepatoma requiring radiotherapy

SUMMARY:
Hepatocellular carcinoma (HCC) is a common cause of cancer mortality in Asia. Most patients were presented with advanced disease. Percutaneous ethanol injection, radiofrequency ablation, and transcatheter arterial chemoembolization (TACE) are not considered as a curative treatment and have achieved very limited success in eradicating large HCC or tumors causing portal vein thrombosis. With the development of novel radiotherapy (RT) technique, RT can be safely given to patients with larger tumor or portal vein thrombosis. However, RT could achieve a tumor response rate of approximately 50 %. Currently, there was a paucity of studies regarding a quantitative biomarker to predict tumor response or forecast the outcome in advance. To optimize the therapeutic index, there is a need to seek effective biomarkers for personal medicine because pretreatment AFP is not always useful as a surrogate marker in some of the patients.

The present study is to investigate whether circulating tumor cell genome in peripheral blood can be used to predict RT response in HCC. We will use the blood sample from patients with locally advanced HCC receiving RT. By using next generation sequencing, We are going to explore the quantity and quality changes of DNAs and RNAs in the patient's serum or plasma. By this way, genomic expression in peripheral blood may play a key role in determining the optimal therapeutic strategies for HCC patients by predicting tumor response to RT.

DETAILED DESCRIPTION:
Patients with hepatocellular carcinoma requiring radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable hepatoma with transarterial chemoembolization (TACE) failure or who are not suitable for TACE. A maximal tumor diameter > 3.0 cm
* Age > 20, and < 80 years
* ECOG 0 or 1
* Life expectancy of at least 12 weeks
* Child-Pugh A
* Cancer of the Liver Italian Program (CLIP) score ≦ 3
* Pretreatment liver function test and renal function test:Total bilirubin < 1.5 times the upper limit of normal (ULN), GOP/GPT ≦ 5 X of upper limit of normal range, Alkaline phosphatase ≦ 4X of ULN, Prothrombin time / partial prothrombin time < 1.5 X of ULN, Serum Creatinine ≦ 1.0 x ULN
* Pretreatment blood count:Hemoglobulin ≧ 9 g/dl, Absolute neutrophil count ≧ 1500/mm3,Platelet count ≧ 100,000/mm3
* Subjects with at least one uni-dimensional or bi-dimensional measurable lesion and lesion must be measured by CT scan

Exclusion Criteria:

* Child-Pugh C
* CLIP score ≧ 4
* Patients with evidence of extrahepatic or metastatic disease
* Patients with evidence of massive ascites
* Patients receiving previous irradiation to liver

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with advanced hepatoma requiring radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Response rate | one month
  The correlation between response rate and circulating tumor cell genome

SECONDARY OUTCOMES:
Overall survival, relapse-free survival | two year

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Wen Chen, MD, Study Director — China Medical University Hosptal
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan